CLINICAL TRIAL: NCT02803112
Title: Pre-hospital and Intra-hospital Temporal Delays in Patients Requiring Emergent Trauma Craniotomy. A 6-year Retrospective Analysis in a Level 1 Trauma Center
Brief Title: Pre-hospital and Intra-hospital Temporal Delays in Patients Requiring Emergent Trauma Craniotomy
Status: Terminated | Type: Observational
Why Stopped: Inactive
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S59232
Record Dates: First submitted 2016-06-06; First posted 2016-06-16 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2016-06

CONDITIONS: Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Emergent craniotomy for traumatic brain injury — Emergent craniotomy for traumatic brain injury (either for removal of an epidural hematoma, subdural hematoma, intraparenchymal hematoma or decompressive craniectomy).

SUMMARY:
The investigators aim to retrospectively map the delays in the acute care of traumatic brain injury patients necessitating emergent craniotomies.

DETAILED DESCRIPTION:
Despite the high incidence of traumatic brain injury (TBI) and the high numbers of emergent craniotomies for TBI performed worldwide, publications reporting on temporal delays in these patients are very scarce. To the best of the investigators' knowledge, there are only 3 publications providing data on the intra-hospital delay and no publications on pre-hospital delay specifically for TBI patients undergoing emergent craniotomies.

The aim of the present study is to retrospectively map delays between the emergency call of the national emergency telephone dispatch to the hospital's medical emergency service (EC) and the surgical skin incision in emergent TBI craniotomies in the investigators' level 1 trauma center and to propose possible measures to improve performance.

ELIGIBILITY:
Inclusion Criteria:

* every patient undergoing 1 of 3 surgical procedures ('removal of epidural hematoma'; 'removal of acute subdural hematoma'; and 'decompressive craniectomy'), performed between February 1, 2010 and January 31, 2016, as recorded in the surgical database of our institution.

Exclusion Criteria:

* who had a delayed clinical or radiological deterioration as a surgical indication;
* who did not have traumatic brain injury as the origin of the intracranial abnormalities;
* in whom not all aforementioned temporal or clinical data were readily available from the electronic patient file; and/or
* who were not admitted via our emergency department.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Traumatic brain injury patients undergoing an emergent craniotomy at our institution (a tertiary referral academic teaching hospital in Leuven, Belgium).
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2010-02; Primary Completion 2016-01 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
Temporal delay between emergency call and the surgical skin incision. | From the trauma onset until 24 hours after the trauma onset.
  Temporal delay (in minutes) between emergency call of the national emergency telephone dispatch to the hospital's medical emergency service and the surgical skin incision during the emergent craniotomy for traumatic brain injury.

SECONDARY OUTCOMES:
Temporal delay between emergency call and arrival at our emergency department. | From the trauma onset until 24 hours after the trauma onset.
  Temporal delay (in minutes) between emergency call of the national emergency telephone dispatch to the hospital's medical emergency service and the arrival at the emergency department of our institution.
Temporal delay between arrival at our emergency department and acquisition of the first head CT slice. | From the trauma onset until 24 hours after the trauma onset.
  Temporal delay (in minutes) between the arrival at the emergency department of our institution and the acquisition of the first head CT slice.
Temporal delay between acquisition of the first head CT slice and arrival in the operating room. | From the trauma onset until 24 hours after the trauma onset.
  Temporal delay (in minutes) between the acquisition of the first head CT slice and arrival in the operating room for emergent trauma craniotomy.
Glasgow Outcome Scale | 6 months after the trauma
  Glasgow Outcome Scale, acquired by a telephone questionnaire, at 6 months after the trauma

CONTACTS AND LOCATIONS:
Overall Officials: Bart Depreitere, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven

IPD SHARING:
Plan to Share IPD: No